CLINICAL TRIAL: NCT06547502
Title: The Study of Pharmacokinetics and Safety of a Single Dose of GZR4 Injection in Subjects with Mild to Moderate Renal Impairment and Subjects with Normal Renal Function
Brief Title: Pharmacokinetics and Safety Profile of a Single Dose GZR4 in Subjects with Renal Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gan and Lee Pharmaceuticals, USA (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GZR4-T2D-104
Record Dates: First submitted 2024-08-07; First posted 2024-08-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Diabetes
Keywords: GZR4; kidney
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Normal renal function (Experimental): GFR between 90-130 ml/min
  Interventions: Drug: GZR4
- Mildly decreased renal function (Experimental): GFR between 60-90 ml/min
  Interventions: Drug: GZR4
- moderately decreased renal function (Experimental): GFR between 30-60 ml/min
  Interventions: Drug: GZR4

INTERVENTIONS:
Drug: GZR4 — single dose

SUMMARY:
This study will be conducted to investigated the effect of decreased kidney function on PK and safety of GZR4 and to guide dosing recommendations in people with kidney impairment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18-75 years (both inclusive) at the time of signing informed consent
* Meeting the pre-defined Glomerular Filtration Rate (GFR) values

Exclusion Criteria:

* Known or suspected hypersensitivity to trial product
* Drugs known to affect creatinine clearance including cimetidine within 14 days or 5 half-lives prior to the day of dosing of GZR4 and during this trial
* Individuals who routinely undergo dialysis or have a history of renal transplantation, hepatorenal syndrome, or acute kidney injury

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2024-07-03 (Actual); Primary Completion 2024-08-20 (Actual); Study Completion 2024-09-05 (Actual)

PRIMARY OUTCOMES:
AUC0-inf | Day1-Day29
AUC0-last | Day1-Day29
Cmax | Day1-Day29

SECONDARY OUTCOMES:
Incidence of TEAE | Day1-Day29
AUC0-168h | Day1-Day29
Tmax | Day1-Day29
T1/2 | Day1-Day29

CONTACTS AND LOCATIONS:
Locations (1):
- Site 1, Suzhou, Jiangsu, China